CLINICAL TRIAL: NCT04991558
Title: Prospective, Single-center Observational Study to Assess the Feasibility and Evaluate the Effectiveness of a Coordinated Healthcare Circuit Dedicated to Patients With Mental and Physical Disabilities Undergoing Planned Surgery
Brief Title: Feasibility and Effectiveness of a Coordinated Healthcare Circuit Dedicated to Patients With Handicap
Acronym: INFRA
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Mutualiste de Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/09-ERA-GHMG
Record Dates: First submitted 2020-12-29; First posted 2021-08-05 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Disabilities Physical; Disabilities Mental

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
France currently has more than 10 million disabled people, including 3 millions who could be better treated. In fact, people with disabilities face many obstacles in accessing care and receiving appropriate support (physical access to certain locations, communication...). Difficulties are also encountered by the healthcare staff, leading to often heterogeneous practices in health establishments.

The INFRA health circuit has been set up at the "Groupe Hospitalier Mutualiste de Grenoble" since June 2018 according to the guidelines published by the French High Authority for Health (HAS) on improving professional practices "Reception, support and organization of care in health establishments for people in situation of handicap "of July 2017. The INFRA nurse collects and anticipates the necessary adaptations for the patient's stay, in conjunction with their caregivers (whether family or institutional). They are an interface with other healthcare professionals to adapt care procedures and protocols (body care, feeding methods, pain management, drug management) to the patient's disability. Before hospitalization and until the patient is discharged, the INFRA nurse transmits to the personnel involved all the information necessary for the proper continuation of care. In addition to legal and regulatory obligations, the INFRA nurse ensures the effective accessibility of the establishment's facilities and premises, and helps maintaining patient autonomy.

The INFRA study is an observational study aimed at assessing the feasibility of the INFRA health circuit and evaluating the benefit for the patients and the healthcare staff.

ELIGIBILITY:
Inclusion Criteria:

* 13 years old or more
* Physical or mental disability, according to french law n°2005-102 of February 11th, 2005
* Requiring an adaptation of the healthcare circuit
* Indication of a planned surgical procedure

Exclusion Criteria:

* Outpatient
* Emergency surgery

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with physical or mental disability, planned for surgical procedure and requiring an adaptation of their healthcare circuit
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who followed the entirety of INFRA circuit | At discharge, assessed up to 4 weeks

SECONDARY OUTCOMES:
Type of pain evaluation scale selected by the INFRA nurse | enrollment
Number of healthcare adaptations implemented during hospitalization | At discharge, assessed up to 4 weeks
Satisfaction of patients and caregivers | At discharge, assessed up to 4 weeks
  Satisfaction survey answered by patients and caregivers
Satisfaction of healthcare staff | At discharge, assessed up to 4 weeks
  Satisfaction survey answered by healthcare staff

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Mutualiste de Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No